CLINICAL TRIAL: NCT04238988
Title: Phase II Study on Carboplatin-Paclitaxel-Pembrolizumab in Neoadjuvant Treatment of Locally Advanced Cervical Cancer
Brief Title: Carboplatin-Paclitaxel-Pembrolizumab in Neoadjuvant Treatment of Locally Advanced Cervical Cancer
Acronym: MITO CERV 3
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2586
Record Dates: First submitted 2019-12-27; First posted 2020-01-23 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Locally Advanced Cervical Cancer
MeSH Terms: interventions — pembrolizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Single arm multicenter phase II trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carboplatin-Paclitaxel-Pembrolizumab (Experimental): Patients will be treated with 3 cycles of neoadjuvant Carboplatin-Paclitaxel chemotherapy (Carboplatin AUC 5 d1 q 21+ Paclitaxel 175 mg/mq d1 q 21)+ Pembrolizumab (200 mg flat dose every 3 weeks).
  After 3 cycles of neo-adjuvant platinum-based chemotherapy patients non progressing will undergo radical surgery.
  After surgery, patients presenting with high risk factors will receive 3 cycles of adjuvant Carboplatin-Paclitaxel chemotherapy + Pembrolizumab in combination and maintenance with Pembrolizumab 200 mg every 3 weeks until progression or unacceptable toxicity or patient consent withdrawal for up to 35 cycles.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Taxol

INTERVENTIONS:
Drug: Pembrolizumab — Humanized antibody used in cancer immunotherapy. It targets the programmed cell death protein 1 (PD-1) receptor of lymphocytes.
  Other Names: Keytruda
Drug: Carboplatin — Chemotherapy medication
Drug: Taxol — Chemotherapy medication
  Other Names: Paclitaxel

SUMMARY:
Single arm multicenter phase II trial evaluating the role of Pembrolizumab in combination to Carboplatin-Paclitaxel chemotherapy in locally advanced cervical cancer patients.

DETAILED DESCRIPTION:
Patients with stage IB2-IIB cervical cancer will be treated with 3 cycles of neoadjuvant Carboplatin-Paclitaxel chemotherapy (Carboplatin AUC 5 d1 q 21+ Paclitaxel 175 mg/mq d1 q 21)+ Pembrolizumab (200 mg flat dose every 3 weeks).

After 3 cycles of neo-adjuvant platinum-based chemotherapy patients non progressing will undergo radical surgery.

After surgery, patients presenting with high risk factors (positive lymphnodes, positive parametria, positive surgical margins or at least 2 of the following risk factor between tumor diameter >3 cm, LVSI, stromal infiltration >1/3) will receive 3 cycles of adjuvant Carboplatin-Paclitaxel chemotherapy + Pembrolizumab in combination and maintenance with Pembrolizumab 200 mg every 3 weeks until progression or unacceptable toxicity or patient consent withdrawal for up to 35 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of FIGO Stage IB2-IIB cervical cancer will be enrolled in this study. Squamous, adenocarcinoma and adenosquamous histotypes are admitted.
2. PDL1+>1% of cell by IHC evaluation in tumor cells
3. Eligible for carboplatin and paclitaxel chemotherapy in accordance with local standards of care
4. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 4 months after the end of treatment
5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
6. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.

   Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of treatment initiation.
9. Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study treatment.
10. No previous systemic chemotherapy or radiation therapy for cervical cancer

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment initiation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior radiotherapy within 2 weeks of start of study treatment for palliative intent. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
4. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
5. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
6. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
8. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
9. Has severe hypersensitivity (≥Grade 3) to Pembrolizumab and/or any of its excipients.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a known history of Human Immunodeficiency Virus (HIV).
14. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection.
15. Has a known history of active TB (Bacillus Tuberculosis).
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
19. History of cerebrovascular accident, pulmonary embolism or untreated grade 3 deep venous thrombosis (DVT) within the past 6 months
20. NCI CTCAE (version 5.0) grade ≥2 enteritis
21. History of myocardial infarction, unstable angina, subarachnoid haemorrhage, stroke or transient ischaemic attack within 6 months before first dose of study drug
22. Clinically significant active cardiovascular disease (e.g., New York Heart Association class II or greater congestive heart failure [CHF], aortic aneurysm)
23. Serious cardiac arrhythmia requiring medication. This does not include asymptomatic atrial fibrillation with controlled ventricular rate
24. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months before study enrolment
25. Pre-existing NCI CTCAE (version 5.0) grade ≥2 peripheral neuropathy

    -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
2-years Progression-free survival | 42 months
  The combination of Pembrolizumab-chemotherapy is expected to increase 2-years progression free survival with respect to historical controls.

SECONDARY OUTCOMES:
Overall survival | 42 months
  The combination of pembrolizumab- chemotherapy is expected to increase overall survival with respect to historical controls
Clinical Response rate | 42 months
  The combination of pembrolizumab-chemotherapy is expected to increase clinical response rate with respect to historical controls
Pathologic optimal response | 42 months
  The combination of pembrolizumab-chemotherapy is expected to increase pathologic response rate with respect to historical controls
Adverse events | 42 months
  The combination of pembrolizumab-chemotherapy is expected to have an acceptable toxicity profile
Quality of life | 42 months
  At baseline, every 3 cycles during the chemotherapy treatment phase, at chemotherapy completion, 6 months after chemotherapy completion, 1 and 2 years after chemotherapy completion and at progression, will be assessed the quality of life of patients according to the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 and CX24. The questionnaires record in a scale from 1 (better outcome) to 4 (worse outcome) the physical, role, emotional, cognitive and social function of patients.
Immune-related gene signatures associated with response or resistance to immune checkpoint blockade | 42 months
  1)Messenger RNA (mRNA) transcript profiling will be performed.
Immune-related gene signatures associated with response or resistance to immune checkpoint blockade | 42 months
  blood sample will be collected before cycle 1, before cycle 6 and at progression. CD3 cells will be isolated and CD4/CD8 ratio will be evaluated by FACS analyses.
Immune-related gene signatures associated with response or resistance to immune checkpoint blockade | 42 months
  serum levels of IL -2, IL-10; TGF- Beta and IL-6 will be assessed.
Immune-related gene signatures associated with response or resistance to immune checkpoint blockade | 42 months
  tumor biopsies at progression will be collected in order to determine the PD-1R infiltrating lymphocyte population before and after treatment.
Immune-related gene signatures associated with response or resistance to immune checkpoint blockade | 42 months
  single and dual staining IHC analysis of: OX40-OX40L; ICOS; PD1, PD-L1, PD2, PDL2 and CTLA-4; FOXP3 and CD4; CD95 and CD95L

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No